CLINICAL TRIAL: NCT00952822
Title: A Phase 1, Prospective, Randomized, Crossover Study to Compare the Pharmacokinetics and Safety of rAHF-PFM Reconstituted in 2 mL Versus 5 mL SWFI in Previously Treated Severe Hemophilia A Patients
Brief Title: Pharmacokinetic Study of ADVATE Reconstituted in 2 mL Sterile Water for Injection
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Baxalta now part of Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 060702
Record Dates: First submitted 2009-08-04; First posted 2009-08-06 (Estimated); Results first posted 2011-07-21 (Estimated); Last update posted 2021-05-24 (Actual); Status verified 2021-04

CONDITIONS: Hemophilia A
MeSH Terms: conditions — Hemophilia A | interventions — Factor VIII

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): ADVATE reconstituted in 2 mL sterile water for infusion
  Interventions: Biological: Antihemophilic factor, recombinant, manufactured protein-free (rAHF-PFM). (Antihemophilic factor is also known as Factor VIII)
- 2 (Active Comparator): ADVATE reconstituted in 5 mL sterile water for infusion
  Interventions: Biological: Antihemophilic factor, recombinant, manufactured protein-free (rAHF-PFM). (Antihemophilic factor is also known as Factor VIII)

INTERVENTIONS:
Biological: Antihemophilic factor, recombinant, manufactured protein-free (rAHF-PFM). (Antihemophilic factor is also known as Factor VIII) — Subjects are randomized to receive an infusion of rAHF-PFM reconstituted in 2 mL sterile water for infusion (SWFI) followed (after a wash-out period) by rAHF-PFM reconstituted in 5 mL SWFI or in 5 mL then 2 mL SWFI(cross-over design). Each subject will receive 2 infusions.
  Other Names: ADVATE

SUMMARY:
The purpose of this study is to determine the pharmacokinetics and safety of Antihemophilic factor, recombinant, manufactured protein-free (rAHF-PFM) reconstituted in 2 mL sterile water for injection (SWFI) and compare with those of rAHF-PFM reconstituted in 5 mL of SWFI.

ELIGIBILITY:
Inclusion Criteria:

* The subject or subject's legally authorized representative has provided written informed consent
* The subject has severe hemophilia A as defined by a baseline FVIII activity <= 1% of normal; tested at screening
* The adolescent/adult subject has a documented history of at least 150 exposure days to FVIII concentrates (either plasma-derived or recombinant), and the pediatric subject has at least 50 exposure days
* The subject is >= 12 to <= 65 years of age for the complete pharmacokinetic assessment and >= 2 to < 12 years for the incremental recovery assessment The subject has a Karnofsky performance score > 60
* The subject is human immunodeficiency virus negative (HIV-) or HIV+ with stable CD4 count >= 200 cells/mm³ (CD4 count determined at screening, if necessary)

Exclusion Criteria:

* The subject has a known hypersensitivity to mouse or hamster proteins or to FVIII concentrates
* The subject has a history of FVIII inhibitors with titer >= 0. 5 BU (Bethesda Assay) or >= 0.4 BU (Nijmegen modification of the Bethesda Assay) any time prior to screening
* The subject has a detectable FVIII inhibitor at screening, >= 0.4 BU (Nijmegen modification of the Bethesda Assay), in the central laboratory
* The subject has severe chronic liver disease as evidenced by, but not limited to, any of the following: International Normalized Ratio (INR) > 1.4, hypoalbuminemia, portal vein hypertension including presence of otherwise unexplained splenomegaly and history of esophageal varices
* The subject has been diagnosed with an inherited or acquired hemostatic defect other than hemophilia A (e.g. qualitative platelet defect or Von Willebrand Disease)
* The subject has received another investigational product within 30 days of enrollment
* The subject's clinical condition may require major or moderate surgery (estimated blood loss > 500 mL) during the period of participation in the study
* Subjects with clinically significant medical, psychiatric, or cognitive illness, or recreational drug/alcohol use that, in the opinion of the investigator, would affect subject safety or compliance
* The subject is a female of childbearing potential with a positive pregnancy test at screening

Ages: 2 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2008-08-08 (Actual); Primary Completion 2009-10-23 (Actual); Study Completion 2009-10-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (11):
- United States (11):
  - Washington D.C., District of Columbia
  - Atlanta, Georgia
  - Lexington, Kentucky
  - Louisville, Kentucky
  - Detroit, Michigan
  - New Brunswick, New Jersey
  - New York, New York
  - Cincinnati, Ohio
  - Portland, Oregon
  - Philadelphia, Pennsylvania
  - Houston, Texas

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment was conducted in the United States at 11 sites. Two cohorts were recruited (adolescent/adults aged ≥12 to ≤65 years and pediatrics aged ≥2 to <12 years).
Pre-assignment Details: Subjects meeting inclusion criteria were randomly assigned to receive a single sequence of 2 pharmacokinetic (PK) infusions of rAHF-PFM: reconstituted in 2mL then 5mL sterile water for injection (SWFI) or vice versa. Before each PK evaluation ≥3 day washout and negative factor VIII inhibitor titer was required. Ten subjects were screen failures
Groups:
- Adolescents/Adults - 2 mL Then 5 mL: Adolescents/Adults - 2 mL then 5 mL: Participants aged ≥12 to ≤65 years who received rAHF-PFM reconstituted in 2 mL SWFI for the 1st Pharmacokinetic (PK) Evaluation, then rAHF-PFM reconstituted in 5 mL SWFI for the 2nd PK Evaluation.
- Adolescents/Adults - 5 mL Then 2 mL: Adolescents/Adults - 5 mL then 2 mL: Participants aged ≥12 to ≤65 years who received rAHF-PFM reconstituted in 5 mL SWFI for the 1st Pharmacokinetic (PK) Evaluation, then rAHF-PFM reconstituted in 2 mL SWFI for the 2nd PK Evaluation.
- Pediatrics - 2 mL Then 5 mL: Pediatrics - 2 mL then 5 mL: Participants aged ≥2 to <12 years who received rAHF-PFM reconstituted in 2 mL SWFI for the 1st Pharmacokinetic (PK) Evaluation, then rAHF-PFM reconstituted in 5 mL SWFI for the 2nd PK Evaluation.
- Pediatrics - 5 mL Then 2 mL: Pediatrics - 5 mL then 2 mL: Participants aged ≥2 to <12 years who received rAHF-PFM reconstituted in 5 mL SWFI for the 1st Pharmacokinetic (PK) Evaluation, then rAHF-PFM reconstituted in 2 mL SWFI for the 2nd PK Evaluation.
Period: 1st Pharmacokinetic Evaluation
Arm/Group | Adolescents/Adults - 2 mL Then 5 mL | Adolescents/Adults - 5 mL Then 2 mL | Pediatrics - 2 mL Then 5 mL | Pediatrics - 5 mL Then 2 mL
Started | 9 | 18 | 11 | 4
Completed | 9 | 17 | 11 | 4
Not Completed | 0 | 1 | 0 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0
Period: 2nd Pharmacokinetic Evaluation
Arm/Group | Adolescents/Adults - 2 mL Then 5 mL | Adolescents/Adults - 5 mL Then 2 mL | Pediatrics - 2 mL Then 5 mL | Pediatrics - 5 mL Then 2 mL
Started | 9 | 17 | 11 | 4
Completed | 9 | 17 | 10 | 4
Not Completed | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Treated Participants: Participants who received at least 1 infusion
Arm/Group | Treated Participants
Number analyzed (Participants) | 42
Age, Continuous [Mean (Standard Deviation); unit: years]
  Pediatrics | 6 (3)
  Adolescents/Adults | 26 (10)
Age, Customized [Count of Participants; unit: Participants]
  ≥2 to <12 years (Number Pediatrics) | 15
  ≥12 to <16 years (Number Adolescents) | 3
  ≥16 to 65 years (Number Adults) | 24
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 42
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 42

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Curve
Description: Area under the factor VIII (FVIII) plasma concentration versus time curve (AUC) from 0 to 48 hours estimated using the linear trapezoidal method
Time Frame: Pharmacokinetic evaluations: 30 minutes pre-infusion up to 48 hours post-infusion
Population: Number of complete crossover participants (per protocol) who received the assigned sequence of 2 infusions: reconstituted in 2mL then 5mL SWFI or in 5mL then 2mL SWFI.
Measure: Geometric Mean (Standard Deviation); unit: IU*h/dL
Groups:
- Adolescents/Adults - 2 mL: Participants aged ≥12 to ≤65 years who received rAHF-PFM reconstituted in 2 mL SWFI
- Adolescents/Adults - 5 mL: Participants aged ≥12 to ≤65 years who received rAHF-PFM reconstituted in 5 mL SWFI
Arm/Group | Adolescents/Adults - 2 mL | Adolescents/Adults - 5 mL
Number analyzed (Participants) | 19 | 19
IU*h/dL | 1257.20 (380.60) | 1297.42 (487.57)
Statistical Analysis 1: Comparison: Adolescents/Adults - 2 mL vs Adolescents/Adults - 5 mL; Test type: Non-Inferiority or Equivalence — Bioequivalence limits of -0.223 to 0.223 in accordance with FDA Guidance for Industry: Statistical Approaches to Establishing Bioequivalence; 2001; Difference of Least-Squares Means = -0.052, 90% CI [-0.117 to 0.012]

2. Secondary Outcome: Total Area Under the Curve
Description: Total AUC when the concentration is extrapolated to zero using the slope of the β-phase of the model
Time Frame: Pharmacokinetic evaluations: 30 minutes pre-infusion up to 48 hours post-infusion
Population: Number of complete crossover participants (intent to treat) who received the assigned sequence of 2 infusions: reconstituted in 2mL then 5mL SWFI or in 5mL then 2mL SWFI.
Measure: Geometric Mean (Standard Deviation); unit: IU*h/dL
Arm/Group | Adolescents/Adults - 2 mL | Adolescents/Adults - 5 mL
Number analyzed (Participants) | 25 | 25
IU*h/dL | 1357.60 (436.24) | 1368.12 (553.21)
Statistical Analysis 1: Comparison: Adolescents/Adults - 2 mL vs Adolescents/Adults - 5 mL; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Difference of Least-Squares Means = -0.016, 90% CI [-0.076 to 0.043]

3. Secondary Outcome: Adjusted in Vivo Incremental Recovery
Description: Increase in factor VIII concentration from pre- to post-infusion
Time Frame: Pharmacokinetic evaluations: 30 minutes pre-infusion to 30 minutes post-infusion
Population: Intent to Treat
Measure: Geometric Mean (Standard Deviation); unit: IU/dL:IU/kg
Groups:
- Pediatrics - 2 mL: Participants aged ≥2 to <12 years who received rAHF-PFM reconstituted in 2 mL SWFI
- Pediatrics - 5 mL: Participants aged ≥2 to <12 years who received rAHF-PFM reconstituted in 5 mL SWFI
Arm/Group | Adolescents/Adults - 2 mL | Adolescents/Adults - 5 mL | Pediatrics - 2 mL | Pediatrics - 5 mL
Number analyzed (Participants) | 26 | 26 | 15 | 14
IU/dL:IU/kg | 1.87 (0.34) | 1.88 (0.40) | 1.33 (0.36) | 1.66 (0.25)

4. Secondary Outcome: Terminal Half-life
Description: Computed from the regression slope in the terminal phase of the model. Terminal half life is the time it takes for the plasma concentration or the amount of drug in the body to be reduced by 50%.
Time Frame: Pharmacokinetic evaluations: 30 minutes pre-infusion up to 48 hours post-infusion
Population: Per Protocol
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Adolescents/Adults - 2 mL | Adolescents/Adults - 5 mL
Number analyzed (Participants) | 19 | 19
hours | 12.54 (3.80) | 12.50 (2.89)

5. Secondary Outcome: Weight-Adjusted Clearance
Description: Computed as the weight-adjusted dose divided by total AUC
Time Frame: Pharmacokinetic evaluations: 30 minutes pre-infusion up to 48 hours post-infusion
Population: Per Protocol
Measure: Mean (Standard Deviation); unit: mL/(kg*h)
Arm/Group | Adolescents/Adults - 2 mL | Adolescents/Adults - 5 mL
Number analyzed (Participants) | 19 | 19
mL/(kg*h) | 3.85 (0.95) | 3.81 (1.20)

6. Secondary Outcome: Mean Residence Time
Description: Computed as total area under the moment curve divided by the total AUC. Total area under the first moment curve (AUMC) estimated by linear trapezoidal methods
Time Frame: Pharmacokinetic evaluations: 30 minutes pre-infusion up to 48 hours post-infusion
Population: Per Protocol
Measure: Mean (Standard Deviation); unit: hours (h)
Arm/Group | Adolescents/Adults - 2 mL | Adolescents/Adults - 5 mL
Number analyzed (Participants) | 19 | 19
hours (h) | 14.79 (5.24) | 14.34 (4.27)

7. Secondary Outcome: Volume of Distribution at Steady State
Description: Computed as weight-adjusted clearance * mean residence time
Time Frame: Pharmacokinetic evaluations: 30 minutes pre-infusion up to 48 hours post-infusion
Population: Per Protocol
Measure: Mean (Standard Deviation); unit: dL/kg
Arm/Group | Adolescents/Adults - 2 mL | Adolescents/Adults - 5 mL
Number analyzed (Participants) | 19 | 19
dL/kg | 0.54 (0.13) | 0.51 (0.13)

8. Secondary Outcome: Maximum Plasma Concentration
Description: Maximal factor VIII concentration post-infusion
Time Frame: Pharmacokinetic evaluations: 30 minutes pre-infusion up to 48 hours post-infusion
Population: Per Protocol
Measure: Geometric Mean (Standard Deviation); unit: IU/dL
Arm/Group | Adolescents/Adults - 2 mL | Adolescents/Adults - 5 mL
Number analyzed (Participants) | 19 | 19
IU/dL | 102.77 (19.35) | 106.46 (17.95)

9. Secondary Outcome: Number and Severity of Infusion Site Reactions
Description: Infusion-related local reactions (including pain, tenderness, erythema, induration, and bruising) and severity were evaluated according to an FDA-defined grading scale (FDA Guidance for Industry: Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers Enrolled in Preventive Vaccine Clinical Trials; 2007).
Time Frame: Within 5 minutes pre-infusion up to 24 hours post-infusion
Population: Participants who received at least 1 infusion
Measure: Number; unit: Participants
Arm/Group | Adolescents/Adults - 2 mL | Adolescents/Adults - 5 mL | Pediatrics - 2 mL | Pediatrics - 5 mL
Number analyzed (Participants) | 27 | 27 | 15 | 15
Participants
  Pain- Mild (Grade 1) | 0 | 0 | 0 | 0
  Pain- Moderate (Grade 2) | 0 | 0 | 0 | 0
  Pain- Severe (Grade 3) | 0 | 0 | 0 | 0
  Pain- Potentially Life Threatening (Grade 4) | 0 | 0 | 0 | 0
  Tenderness- Mild (Grade 1) | 0 | 0 | 0 | 0
  Tenderness- Moderate (Grade 2) | 0 | 0 | 0 | 0
  Tenderness- Severe (Grade 3) | 0 | 0 | 0 | 0
  Tenderness- Potentially Life Threatening (Grade 4) | 0 | 0 | 0 | 0
  Erythema- Mild (Grade 1) | 0 | 0 | 0 | 0
  Erythema- Moderate (Grade 2) | 0 | 0 | 0 | 0
  Erythema- Severe (Grade 3) | 0 | 0 | 0 | 0
  Erythema- Potentially Life Threatening (Grade 4) | 0 | 0 | 0 | 0
  Induration- Mild (Grade 1) | 0 | 0 | 1 | 0
  Induration- Moderate (Grade 2) | 0 | 0 | 0 | 0
  Induration- Severe (Grade 3) | 0 | 0 | 0 | 0
  Induration- Potentially Life Threatening (Grade 4) | 0 | 0 | 0 | 0
  Bruising- Mild (Grade 1) | 0 | 0 | 1 | 0
  Bruising- Moderate (Grade 2) | 0 | 0 | 0 | 0
  Bruising- Severe (Grade 3) | 0 | 0 | 0 | 0
  Bruising- Potentially Life Threatening (Grade 4) | 0 | 0 | 0 | 0

10. Secondary Outcome: Infusion Site Pain
Description: Pain was assessed by participants (≥5 years of age) on a visual analog scale (VAS) from 0 (no pain) to 100 (worst possible pain).
Time Frame: Within 5 minutes post-infusion up to 24 hours post-infusion
Population: Participants who received at least 1 infusion
Measure: Median (Full Range); unit: Scores on a scale
Groups:
- Adolescents/Adults - 5 mL: Participants aged ≥12 to ≤65 years who received rAHF-PFM reconstituted in 5 mL SWFI (note: 24 hours after infusion n=26)
- Pediatrics at Least 5 Years of Age - 2 mL: Participants aged ≥5 years to <12 years who received rAHF-PFM reconstituted in 2 mL SWFI (note: 6 hours after infusion n=7)
- Pediatrics at Least 5 Years of Age - 5 mL: Participants aged ≥5 years to <12 years who received rAHF-PFM reconstituted in 5 mL SWFI (note: 24 hours after infusion n=7)
Arm/Group | Adolescents/Adults - 2 mL | Adolescents/Adults - 5 mL | Pediatrics at Least 5 Years of Age - 2 mL | Pediatrics at Least 5 Years of Age - 5 mL
Number analyzed (Participants) | 26 | 27 | 8 | 8
Scores on a scale
  Within 5 minutes (immediately) after infusion | 0 [0 to 12] | 0 [0 to 27] | 8 [0 to 37] | 4 [0 to 61]
  60 ± 5 minutes after infusion | 0 [0 to 3] | 0 [0 to 4] | 2.5 [0 to 66] | 1 [0 to 7]
  6 hours ± 30 minutes after infusion | 0 [0 to 3] | 0 [0 to 2] | 0 [0 to 8] | 0 [0 to 4]
  24 hours after infusion | 0 [0 to 2] | 0 [0 to 3] | 0 [0 to 8] | 0 [0 to 2]

ADVERSE EVENTS:
Time Frame: During course of study
Description: AEs were collected by the investigators at study visits, and may result from laboratory and vital sign assessments collected or measured at the study visits
Groups:
- Adolescents/Adults; Pediatrics: Participants aged ≥12 to ≤65 years who received at least one infusion
Arm/Group | Adolescents/Adults | Pediatrics
Serious Adverse Events (participants affected / at risk) | 0/27 | 1/15
Other Adverse Events (participants affected / at risk) | 1/27 | 10/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Adolescents/Adults (N=27) | Pediatrics (N=15)
Pyrexia (General disorders) | 0 (0) | 1 (1) — Not related to study drug
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Adolescents/Adults (N=27) | Pediatrics (N=15)
Allergy to arthropod sting (Immune system disorders) | 0 | 1 (1) — Not related to study drug
Arthropod bite (Injury, poisoning and procedural complications) | 1 (1) | 2 (2) — Not related to study drug
Catheter thrombosis (General disorders) | 0 | 1 (1) — Not related to study drug
Conjunctival hemorrhage (Eye disorders) | 0 | 1 (1) — Not related to study drug
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 5 (5) — Not related to study drug
Ear infection (Infections and infestations) | 0 | 1 (1) — Not related to study drug
Hemarthrosis (Musculoskeletal and connective tissue disorders) | 0 | 1 (1) — Not related to study drug
Injection site hematoma (General disorders) | 0 | 1 (1) — Not related to study drug
Injection site swelling (General disorders) | 0 | 1 (1) — Not related to study drug
Joint range of motion (Musculoskeletal and connective tissue disorders) | 0 | 1 (1) — Not related to study drug

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Baxter's agreements with PIs vary per individual PI, but contain common elements. For this study, PIs are restricted from independently publishing results until the earlier of the primary multicenter publication or 1 year after study completion. Baxter requires a review of results communications (e.g., for confidential information) up to 90 days prior to submission or communication. Baxter may request an additional delay of up to 60 days (e.g., to allow for intellectual property protection).